CLINICAL TRIAL: NCT04472520
Title: Use of AliveCor ECG Monitoring to Replicate ECG Lead Recording
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dan Sorajja, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-002678
Record Dates: First submitted 2020-06-05; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subject getting an ECG (Experimental): Subjects getting an ECG will have AliveCore tracings obtained in 3 configurations; between right hand and left hand, between left hand and left lower leg (thigh, calf, and foot) and between right hand and left lower leg (thigh, calf, and foot).These configurations will be obtained with the participant lying in bed and in a sitting position.
  Interventions: Device: AliveCor Heart Monitor

INTERVENTIONS:
Device: AliveCor Heart Monitor — Records single-channel ECG rhythms

SUMMARY:
The researchers are trying to determine whether the Alivecor device can simulate other electrocardiogram (ECG) leads to record electrical activity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals greater than 18 years old getting an ECG

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram (ECG) QT Interval | 1 day
  The QT interval represents the time of ventricular activity including both depolarization and repolarization. It is measured from the beginning of the QRS complex to the end of the T wave. Normally, the QT interval is 0.36 to 0.44 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Dan Sorajja, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials